CLINICAL TRIAL: NCT06795594
Title: Cheek Acupuncture Therapy Vs. Standard Therapy for Pain Control After Elective Caesarean Section - a Randomized Controlled Trial
Brief Title: Effectiveness of Cheek Acupuncture Therapy for Pain Control After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TREC2024-KY090.R1
Record Dates: First submitted 2024-12-08; First posted 2025-01-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-01

CONDITIONS: Acupuncture Analgesia
Keywords: Cheek acupuncture therapy; Acupuncture; Cesarean delivery; Pain control; Postoperative pain management
MeSH Terms: conditions — Agnosia | interventions — Sufentanil; Ondansetron

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cheek Acupuncture group (Experimental): Each patient in the cheek acupuncture group received cheek acupuncture therapy as a supplement to the postoperative patient-controlled analgesia pump. The selected cheek acupuncture points included four bilateral points for the neck, back, waist, and sacrum, as well as four abdominal holographic points, totaling eight points. Cheek acupuncture procedure: The patient was placed in a supine position, and the acupoint skin was routinely disinfected. Acupuncture needles of 0.15mm by 15mm were used, inserted quickly and vertically to a depth of 10 to 15mm without seeking the sensation of "qi" arrival. The needles were left in place for 30 minutes and then removed, followed by applying a cotton ball to press on the needle holes for a moment. The intervention was conducted twice, each time for 30 minutes, with the first session immediately after completing the anesthesia operation and the second session at 23.5 hours postoperatively.
  Interventions: Procedure: cheek acupuncture; Drug: sufentanil 2 µg/kg + ondansetron 0.2 mg/kg
- Control group (Sham Comparator): The control group used only a patient-controlled analgesia (PCA) pump for postoperative pain relief. The pump contained 2 micrograms per kilogram of sufentanil and 0.2 milligrams per kilogram of ondansetron, with a total volume of 100 milliliters. The pump was set to deliver a continuous infusion of 2 milliliters per hour, with the option for patients to self-administer an additional 2-milliliter bolus dose as needed, with a minimum interval of 15 minutes between doses. If the primary analgesic measures were insufficient to control pain, diclofenac sodium suppositories were provided as rescue analgesia, based on patient needs. The use of these suppositories was based on individual patient pain assessments and the need for additional pain relief.
  Interventions: Drug: sufentanil 2 µg/kg + ondansetron 0.2 mg/kg

INTERVENTIONS:
Procedure: cheek acupuncture — Cheek Acupuncture
  Arms: Cheek Acupuncture group
Drug: sufentanil 2 µg/kg + ondansetron 0.2 mg/kg — The patient-controlled analgesia (PCA) pump held a solution of 2 µg/kg sufentanil and 0.2 mg/kg ondansetron in 100 ml. It infused 2 ml/hour continuously, allowing patients to self-administer an extra 2 ml bolus every 15 minutes if needed. For inadequate pain control, diclofenac sodium suppositories were used as rescue analgesia, depending on individual pain assessments and the requirement for extra relief.

SUMMARY:
This study investigates whether cheek acupuncture therapy can alleviate postoperative pain in cesarean section patients and explores its mechanisms of action through a prospective randomized controlled clinical trial.

DETAILED DESCRIPTION:
Pain control after cesarean delivery, if inadequately managed, can impact the prognosis of the mother and the health of the infant. There is an urgent need to explore safer, more effective, and straightforward non-pharmacological adjunctive interventions to alleviate the pain associated with cesarean section. Cheek acupuncture therapy is a green micro-acupuncture treatment that has shown significant improvement in various types of pain and holds great potential for relieving perioperative pain. To practice the concept of perioperative acupuncture medicine, this study aims to investigate whether cheek acupuncture therapy can alleviate postoperative pain in cesarean section patients and to explore the mechanisms by which it exerts its effects, through a prospective randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are classified as American Society of Anesthesiologists (ASA) physical status I to III.
2. Scheduled for elective cesarean delivery under spinal anesthesia.
3. Patients are aged between 19 to 45 years old.
4. Patients have provided written informed consent.

Exclusion Criteria:

1. Local skin infection at the acupuncture sites in the cheek area.
2. Cases where spinal anesthesia fails and general anesthesia is required.
3. Patients with conditions such as recurrent alcohol abuse, fever, convulsions, or cardiopulmonary failure.
4. Patients who have used opioid medications at least 6 months prior to surgery.
5. Patients who are unable to understand the consent form and study questionnaire, including those with cognitive impairments.
6. Patients with a history of psychiatric illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (0-10) pain score during movement | 24 hours postoperatively, which is half an hour after the completion of the second cheek acupuncture treatment
  Numeric Rating Scale, this scale is a validated tool for measuring pain intensity, with scores ranging from 0 (no pain) to 10 (the most severe pain imaginable).The higher the score, the more severe the pain.

SECONDARY OUTCOMES:
the proportion of patients with NRS pain score ≥ 6 | 24 hours postoperatively, which is half an hour after the completion of the second cheek acupuncture treatment
  Assess the proportion of severe pain by calculating the ratio of NRS pain scores that are greater than or equal to 6.
NRS pain score during movement | morning of the day of discharge (assessed up 7 days)
  Numeric Rating Scale, this scale is a validated tool for measuring pain intensity, with scores ranging from 0 (no pain) to 10 (the most severe pain imaginable).The higher the score, the more severe the pain.
The Hospital Anxiety and Depression Scale (HADS)-A | morning of the day of discharge (assessed up 7 days)
  The Hospital Anxiety and Depression Scale (HADS)-A is a subscale of the HADS, which is a self-assessment questionnaire used to screen for symptoms of anxiety and depression in patients within a non-psychiatric hospital setting. The 'A' stands for Anxiety, and the HADS-A specifically measures the severity of anxiety symptoms. It consists of 7 items rated on a 4-point scale, with scores ranging from 0 to 21, where higher scores indicate greater anxiety.
HADS-D score | morning of the day of discharge (assessed up 7 days)
  The Hospital Anxiety and Depression Scale (HADS)-D is a subscale of the HADS, which is designed to identify anxiety and depression in patients within hospital settings. The 'D' stands for Depression, and this subscale specifically assesses the severity of depressive symptoms. It includes 7 items rated on a 4-point scale, with scores ranging from 0 to 21, where higher scores indicate more severe depressive symptoms.
ISI score | morning of the day of discharge (assessed up 7 days)
  The ISI-(0-28) refers to the Insomnia Severity Index, which is a self-administered questionnaire used to evaluate the severity of insomnia. It consists of 7 items scored on a 5-point Likert scale, ranging from 0 (no difficulty) to 4 (extreme difficulty). The total score ranges from 0 to 28, with higher scores indicating greater severity of insomnia.
QoR15 score | morning of the day of discharge (assessed up 7 days)
  The QoR15 score is a measure used to assess the quality of recovery following surgery. It stands for "Quality of Recovery-15," and it is a 15-item questionnaire that evaluates various aspects of a patient's recovery, such as pain, nausea, vomiting, fatigue, and return to physical and cognitive function. The score ranges from 0 to 150, with a higher score indicating a better quality of recovery.
HCRP | 48 hours postoperatively
  HCRP stands for High-Sensitivity C-Reactive Protein. It is a blood test that measures the levels of C-reactive protein (CRP), which is a marker of inflammation in the body. High-sensitivity CRP tests can detect low levels of CRP, making it a useful tool for monitoring inflammation, cardiovascular risk, and the effectiveness of treatments for various inflammatory conditions.
Beta-endorphin | 48 hours postoperatively
  Beta-endorphin is an endogenous opioid peptide produced by the body, consisting of 31 amino acids. It is a natural painkiller and plays a role in reducing pain and stress. Beta-endorphin is released in response to stress, pain, or the use of opioids, and it contributes to the body's reward system and regulation of mood. It is also associated with the release of adrenaline during stress or intense physical activity.
Postoperative adverse reactions | From date of randomization until the date of discharge, assessed up to 7 days
  Explore whether cheek acupuncture intervention increases postoperative adverse reactions, including dizziness, abdominal bloating, nausea, vomiting, fatigue and so on.
Postoperative severe complications | From date of randomization until the date of discharge, assessed up to 7 days
  Postoperative severe complications, including pulmonary complications, heart failure, liver dysfunction, kidney dysfunction, coagulation function, SIRS (Systemic Inflammatory Response Syndrome), stroke, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No